CLINICAL TRIAL: NCT05915130
Title: A Study Protocol for Testing an Innovative Gait Training Program in Immersive Virtual Reality for Healthy Older Adults
Brief Title: An Innovative Gait Training Program in Immersive Virtual Reality for Healthy Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aix Marseille Université (Other)
Responsible Party: Principal Investigator, Lisa Delbes, Principal investigator, Aix Marseille Université
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GTPVR
Record Dates: First submitted 2023-05-23; First posted 2023-06-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Fall; Elderly
Keywords: adaptive behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality training program (Experimental): In the VR group, participants will practice the training sessions in an experimental room. In one training session, participants will negotiate 60 trials. Participants will practice gait training sessions in a fully immersive virtual reality. They will negotiate virtual obstacles such as avoiding a rock or crossing over a tree root, thus improving their gait adaptability capacities.
  Interventions: Behavioral: Gait training
- Nordic walking training program (Experimental): Participants will be instructed to walk with poles continuously around the park. Each training session will consist of a warm-up (10 min), main exercise (40 min), and cool-down (5 min) periods. Participants will adapt their locomotion to uneven terrain. They will negotiate natural obstacles such as avoiding a rock or crossing over a tree root, thus improving their gait adaptability capacities.
  Interventions: Behavioral: Gait training

INTERVENTIONS:
Behavioral: Gait training — They will negotiate (natural or virtual) obstacles such as avoiding a rock or crossing over a tree root, thus improving their gait adaptability capacities.

SUMMARY:
Background Impaired gait adaptability is one of the major causes of falls among older adults by producing inappropriate gait adjustments in cluttered environments. Training programs designed to improve gait adaptability behavior in a systemic approach may prevent falls in older adults. Recently, the technology of virtual reality has appeared as a relevant gait training tool based on its training implementation potential. The present study was designed to compare the effectiveness of a virtual reality gait training program (VR group) for improving gait adaptability behavior and thus, reducing the risk of falls relative to a conventional training program of Nordic walkway (NW group). We hypothesize that the virtual reality gait training program will lead to greater gait adaptability improvements.

Methods The protocol describes a randomized controlled trial with pre-tests, post-tests, retention tests and follow-up. Forty healthy independent living community dweller participants (65-80 years) will be allocated, after a general medical examination, to the VR or the NW group for a training program of six weeks. Primary outcome related to gait adaptability capacities and acceptance of the virtual reality device will be assessed in pre- and post-intervention and one month after the completion of the training program (retention). A follow-up will be done during the 12 months after the completion of the gait training program.

Discussion This study will demonstrate the relative relevance of a gait training program in virtual reality versus a conventional one for improving gait adaptability behavior in healthy older adults and thus preventing falls.

ELIGIBILITY:
Inclusion Criteria:

* aged between 65 and 80
* with weekly moderate to vigorous physical activity

Exclusion Criteria:

* inability to practice activity at a moderate or vigorous intensity
* moderate or severe cognitive impairments
* severe non-corrected visual impairments
* uncontrolled psychiatric disorders

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Gait adaptability capacities | Pre-intervention (week 1)
  Gait adaptability capacities will be assessed by a specific gait test created to assess gait parameters during goal-directed tasks. Feet positions will be measured by a seven-meter-long portable pressure-sensitive walkway GaitRite® (CIR Systems, Inc., Franklyn, NY, USA) in the real world. Firstly, participants will be instructed to walk at a normal pace on the walkway. The average preferred gait speed, step length, and step duration (with their variabilities) will be calculated over 6 trials. Afterwards, physical obstacles will be placed on the walkway. Participants will perform 3 different locomotor tasks: simple locomotor pointing, crossing-over, and stepping-over tasks (see Figure 4). They will perform 10 trials of each goal-directed task. By recording successive feet positions in relation to the obstacles, gait adaptability behavior will be analyzed through performance, inter-trials and trial-by-trial analyses.
Gait adaptability capacities | Post-intervention (week 8)
  Gait adaptability capacities will be assessed by a specific gait test created to assess gait parameters during goal-directed tasks. Feet positions will be measured by a seven-meter-long portable pressure-sensitive walkway GaitRite® (CIR Systems, Inc., Franklyn, NY, USA) in the real world. Firstly, participants will be instructed to walk at a normal pace on the walkway. The average preferred gait speed, step length, and step duration (with their variabilities) will be calculated over 6 trials. Afterwards, physical obstacles will be placed on the walkway. Participants will perform 3 different locomotor tasks: simple locomotor pointing, crossing-over, and stepping-over tasks (see Figure 4). They will perform 10 trials of each goal-directed task. By recording successive feet positions in relation to the obstacles, gait adaptability behavior will be analyzed through performance, inter-trials and trial-by-trial analyses.
Gait adaptability capacities | Retention (week 12)
  Gait adaptability capacities will be assessed by a specific gait test created to assess gait parameters during goal-directed tasks. Feet positions will be measured by a seven-meter-long portable pressure-sensitive walkway GaitRite® (CIR Systems, Inc., Franklyn, NY, USA) in the real world. Firstly, participants will be instructed to walk at a normal pace on the walkway. The average preferred gait speed, step length, and step duration (with their variabilities) will be calculated over 6 trials. Afterwards, physical obstacles will be placed on the walkway. Participants will perform 3 different locomotor tasks: simple locomotor pointing, crossing-over, and stepping-over tasks (see Figure 4). They will perform 10 trials of each goal-directed task. By recording successive feet positions in relation to the obstacles, gait adaptability behavior will be analyzed through performance, inter-trials and trial-by-trial analyses.
Acceptance of the head-mounted device | Pre-intervention (week 1)
  For the VR group only, VR-HMD acceptance before and after use will be assessed using the Technology Acceptance Model. According to this model, intention to use a technology is positively predicted by its perceived usefulness and its perceived ease of use. VR-HMD acceptance will be assessed through four variables: perceived usefulness, perceived ease of use, perceived enjoyment, and intention to use.
  (12 items with a 1-10 Likert scale; a higher score means a better outcome)
Acceptance of the head-mounted device | Post-intervention (week 8)
  For the VR group only, VR-HMD acceptance before and after use will be assessed using the Technology Acceptance Model. According to this model, intention to use a technology is positively predicted by its perceived usefulness and its perceived ease of use. VR-HMD acceptance will be assessed through four variables: perceived usefulness, perceived ease of use, perceived enjoyment, and intention to use.
  (12 items with a 1-10 Likert scale; a higher score means a better outcome)

SECONDARY OUTCOMES:
Mobility | Pre-intervention (week 1)
  Mobility evaluation will be assessed with the Timed Up-and-Go (TUG) test (performance in s).
Mobility | Post-intervention (week 8)
  Mobility evaluation will be assessed with the Timed Up-and-Go (TUG) test (performance in s).
Mobility | Retention (week 12)
  Mobility evaluation will be assessed with the Timed Up-and-Go (TUG) test (performance in s).
Balance | Pre-intervention (week 1)
  Balance evaluation will be assessed with the Unipedal stance test (performance in s).
Balance | Post-intervention (week 8)
  Balance evaluation will be assessed with the Unipedal stance test (performance in s).
Balance | Retention (week 12)
  Balance evaluation will be assessed with the Unipedal stance test (performance in s).
Motivation | Pre-intervention (week 1)
  Motivation for physical activity will be assessed using the ÉMAPS questionnaire recently validated in French (18 items with a 1-7 Likert scale; a higher score means a better outcome)
Motivation | Post-intervention (week 8)
  Motivation for physical activity will be assessed using the ÉMAPS questionnaire recently validated in French (18 items with a 1-7 Likert scale; a higher score means a better outcome)
Motivation | Retention (week 12)
  Motivation for physical activity will be assessed using the ÉMAPS questionnaire recently validated in French (18 items with a 1-7 Likert scale; a higher score means a better outcome)
Intrinsic motivation | Pre-intervention (week 1)
  Intrinsic motivation will be assessed using the Inventory Motivation inventory (IMI) questionnaire (22 items with a 1-7 Likert scale; a higher score means a better outcome)
Intrinsic motivation | Post-intervention (week 8)
  Intrinsic motivation will be assessed using the Inventory Motivation inventory (IMI) questionnaire (18 items with a 1-7 Likert scale; a higher score means a better outcome)
Intrinsic motivation | Retention (week 12)
  Intrinsic motivation will be assessed using the Inventory Motivation inventory (IMI) questionnaire (18 items with a 1-7 Likert scale; a higher score means a better outcome)
Fear of falling | Pre-intervention (week 1)
  Fear of falling will be assessed using the French version of the Modified-Falls Efficacy Scale (14 items with a 1-10 Likert scale; a higher score means a worse outcome)
Fear of falling | Post-intervention (week 8)
  Fear of falling will be assessed using the French version of the Modified-Falls Efficacy Scale (14 items with a 1-10 Likert scale; a higher score means a worse outcome)
Fear of falling | Retention (week 12)
  Fear of falling will be assessed using the French version of the Modified-Falls Efficacy Scale (14 items with a 1-10 Likert scale; a higher score means a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Movement Sciences, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided